CLINICAL TRIAL: NCT00071526
Title: Urinary Vitamin C Loss in Subjects With and Without Diabetes
Brief Title: Urinary Vitamin C Loss in Diabetic Subjects
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040021; 04-DK-0021
Record Dates: First submitted 2003-10-27; First posted 2003-10-28 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01-23

CONDITIONS: Diabetes
Keywords: Renal Threshold; Diabetes Mellitus; Proteinuria; Plasma Concentrations; Healthy Volunteer
MeSH Terms: conditions — Diabetes Mellitus; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diabetes Type I: Subjects with Type I diabetes mellitus
- Diabetes Type II: Subjects with Type II diabetes mellitus
- Healthy Volunteers: Healthy Volunteers

SUMMARY:
Several studies have reported that diabetic subjects have lower plasma vitamin C concentrations than non-diabetic subjects. Although urinary vitamin C loss in diabetic subjects was reported to be increased in two studies, these are difficult to interpret due to lack of controlled vitamin C intake, inadequate sampling, lack of control subjects, or methodology uncertainties in vitamin C assay and sample processing. Consequently, it is unclear whether diabetic subjects truly have both low plasma and high urine vitamin C concentrations. We propose that low plasma vitamin C concentrations in diabetic subjects are due in part to inappropriate renal loss of vitamin C in these subjects but not in healthy controls. We will study nondiabetic controls and cohorts with diabetes. Vitamin C concentrations in plasma, RBCs, and urine will be measured in outpatients. In those willing to be admitted to the Clinical Center, we will measure vitamin C pharmacokinetics to determine the relative bioavailability for vitamin C in individuals with and without abnormal urinary loss of vitamin C (or renal leak). Single nucleotide polymorphisms (SNPs) will be determined in genomic DNA responsible for the two proteins mediating sodium dependent vitamin C transport, SVCT1 and SVCT2. We will also explore mechanisms underlying abnormal urinary vitamin C loss.

DETAILED DESCRIPTION:
Several studies have reported that diabetic subjects have lower plasma vitamin C concentrations than non-diabetic subjects. Although urinary vitamin C loss in diabetic subjects was reported to be increased in two studies, these are difficult to interpret due to lack of controlled vitamin C intake, inadequate sampling, lack of control subjects, or methodology uncertainties in vitamin C assay and sample processing. Consequently, it is unclear whether diabetic subjects truly have both low plasma and high urine vitamin C concentrations. We propose that low plasma vitamin C concentrations in diabetic subjects are due in part to inappropriate renal loss of vitamin C in these subjects but not in healthy controls. We will study nondiabetic controls and cohorts with diabetes. Vitamin C concentrations in plasma, RBCs, and urine will be measured in outpatients. In those willing to be admitted to the Clinical Center, we will measure vitamin C pharmacokinetics to determine the relative bioavailability for vitamin C in individuals with and without abnormal urinary loss of vitamin C (or renal leak). Single nucleotide polymorphisms (SNPs) will be determined in genomic DNA responsible for the two proteins mediating sodium dependent vitamin C transport, SVCT1 and SVCT2. We will also explore mechanisms underlying abnormal urinary vitamin C loss.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be included in the study, study subjects should be:

* Aged 18-65 years.
* Either:

  * Have no diagnosis of diabetes: "nondiabetic controls", or
  * Have a diagnosis in their medical history of either Type 1 or Type 2 diabetes

EXCLUSION CRITERIA (for outpatient study, arm 1)

Exclusion criteria will include the following:

* Unable or unwilling to provide a signed and dated informed consent form
* Unable or unwilling to comply with study procedures and lifestyle considerations

EXCLUSION CRITERIA (for inpatient studies, arms 2 and 3)

Study participants interested in participating in Arms 2 and/or 3 will be excluded from this further participation if they meet any of the following:

* significant organ malfunction leading to clinical instability including liver disease, pulmonary disease, ischemic heart disease, heart failure, stroke, peripheral vascular disease, and anemia at investigator discretion
* other serious or chronic illness; history of serious or chronic illness; coronary artery disease, or peripheral vascular disease resulting in clinical instability
* pregnancy or lactation
* presence of other conditions which, in the judgment of the investigators, can influence vitamin C metabolism or vitamin C renal handling

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2006-04-11 (Actual)

PRIMARY OUTCOMES:
Plasma, neutrophil and RBC Vitamin C concentrates | end of study
  Measurements of plasma, neutrophil and red blood cell vitamin c concentrations in diabetic subjects as compared to healthy controls.

SECONDARY OUTCOMES:
Urinary vitamin C concentration | end of study
  Measurements of urinary vitamin c concentrations in diabetic subjects as compared to healthy controls.
Determine the renal threshold and relative bioavailability for vitamin C | end of study
  Calculate renal threshold of vitamin C in diabetic subjects as compared to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Ifechukwude C Ebenuwa, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Levine M. New concepts in the biology and biochemistry of ascorbic acid. N Engl J Med. 1986 Apr 3;314(14):892-902. doi: 10.1056/NEJM198604033141407. No abstract available. PMID 3513016
- [Background] Goodwin JS, Goodwin JM, Garry PJ. Association between nutritional status and cognitive functioning in a healthy elderly population. JAMA. 1983 Jun 3;249(21):2917-21. PMID 6842805
- [Background] Fata FT, Herzlich BC, Schiffman G, Ast AL. Impaired antibody responses to pneumococcal polysaccharide in elderly patients with low serum vitamin B12 levels. Ann Intern Med. 1996 Feb 1;124(3):299-304. doi: 10.7326/0003-4819-124-3-199602010-00003. PMID 8554224
- [Derived] Ebenuwa I, Violet PC, Tu H, Lee C, Munyan N, Wang Y, Niyyati M, Patra K, Wilkins KJ, Parrow N, Levine M. Altered RBC deformability in diabetes: clinical characteristics and RBC pathophysiology. Cardiovasc Diabetol. 2024 Oct 18;23(1):370. doi: 10.1186/s12933-024-02453-2. PMID 39425096
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-DK-0021.html